CLINICAL TRIAL: NCT00247754
Title: VP3: Vancouver Primary Prevention Program (Anxiety Disorders Prevention in School Children)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: B01-0072
Record Dates: First submitted 2005-10-31; First posted 2005-11-02 (Estimated); Last update posted 2005-11-02 (Estimated); Status verified 2005-10

CONDITIONS: Anxiety
Keywords: Anxiety; Therapy; Behaviour
MeSH Terms: conditions — Anxiety Disorders; Behavior

INTERVENTIONS:
Behavioral: Cognitive Behaviour Treatment

SUMMARY:
Objective:

1. To evaluate the efficacy of a school-based cognitive behavior therapy (CBT) program in reducing anxiety disorder symptoms in at-risk public school children.
2. To determine whether parent education and involvement improves outcome in anxious children treated with CBT.
3. To determine the ability of school personnel in a) recognizing classroom behaviors as anxiety disordered after targeting training of observable child behaviors e.g., avoidance, over-worry, etc.), and b) delivering a cognitive behavior intervention and
4. To evaluate a new measure of teacher-rated anxiety disorder symptoms in children.

Hypothesis:

1. A CBT oriented intervention as delivered by school personnel will be superior to an attention control procedure in reducing anxiety symptoms in at-risk children.
2. Children who have parental involvement will post stronger and more enduring treatment gains.

ELIGIBILITY:
Inclusion Criteria:

Children enrolled in school between the ages of 7 and 13 who display anxiety symptoms.

1. Anxiety disorder symptoms (identified by a score of 56 or higher on the MASC; and teacher report, and /or parent recommendation) as the primary presenting problem. An enrolled child must have at least 2 of these criterions.
2. Fluency in English.
3. Parent willingness to sign consent form and to complete required assessments.
4. Student willingness to participate (child assent) in 10-week affective education program and completion of required assessments.

Exclusion Criteria:

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 281
Dates: Start 2002-11; Study Completion 2005-06

PRIMARY OUTCOMES:
Anxiety symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Miller, PhD, R.Psych., Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Faculty of Education, Vancouver, British Columbia, Canada